CLINICAL TRIAL: NCT03279263
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Add-on Study of MLR 1023 in Adults With Uncontrolled Type 2 Diabetes on Metformin Therapy
Brief Title: An Add-on Study of MLR-1023 in Adults With Uncontrolled Type 2 Diabetes on Metformin Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Melior Pharmaceuticals (Other)
Collaborators: Bukwang Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BK-MD-202
Record Dates: First submitted 2017-08-25; First posted 2017-09-12 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 5-(3-methylphenoxy)-2(1H)-pyrimidinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MLR-1023 25mg QD (Experimental): MLR-1023 25mg QD Tablet
  Interventions: Drug: MLR-1023
- MLR-1023 50mg QD (Experimental): MLR-1023 50mg QD Tablet
  Interventions: Drug: MLR-1023
- MLR-1023 100mg QD (Experimental): MLR-1023 100mg QD Tablet
  Interventions: Drug: MLR-1023
- Placebo (Placebo Comparator): Placebo QDTablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MLR-1023 — MLR-1023 Tablets
  Arms: MLR-1023 100mg QD; MLR-1023 25mg QD; MLR-1023 50mg QD
Other: Placebo — Matching Placebo Tablets
  Arms: Placebo

SUMMARY:
This Phase 2, multi-center, double-blind, randomized, placebo-controlled, parallel group, add-on study of MLR 1023 in adults with uncontrolled T2DM on metformin anti diabetic monotherapy is designed to evaluate the efficacy and safety of MLR 1023 in combination with metformin in subjects with uncontrolled T2DM.

DETAILED DESCRIPTION:
Medical management of T2DM involves diet, exercise, weight management, and pharmacotherapy. Pharmacological agents, such as metformin, α-glucosidase inhibitors, orlistat, and thiazolidinediones, have been shown to decrease incident diabetes. Metformin has the strongest evidence base and demonstrated long-term safety as pharmacological therapy for diabetes treatment. The American Diabetes association position statement on diabetes care recommends that if Hemoglobin A1C (HbA1C) targets are not achieved after approximately 3 months of metformin anti-diabetic monotherapy, a combination of metformin and one of several oral treatment options should be considered.

In this study, subjects with a diagnosis of T2DM who are not adequately controlled (HbA1C between 7.0% and 10.0%, inclusive) and started metformin therapy at least 3 months prior to Screening will be recruited into the study. Subjects will continue taking metformin for the duration of the study and once daily oral MLR 1023 or placebo will be added to metformin.

The efficacious dose-level range of MLR 1023 in diabetic subjects is anticipated to be between 25 and 100 mg. Therefore, the efficacy, safety, and tolerability of 25 mg and 50 mg doses in addition to the 100 mg dose that was shown to be effective in the Phase 2a proof of concept study will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 75 years, inclusive.
2. Diagnosis of T2DM.
3. Body mass index (BMI) between 20 and 40 kg/m2.
4. HbA1C between 7.0% and 10.0%.
5. Treated with metformin as the only anti-diabetic therapy.
6. Metformin dosage must have been stable and unchanged for at least 3 months prior to Screening and at a dose of at least 1,500 mg/day or the maximum tolerated dose if less than 1,500 mg/day.
7. Able and willing to comply with the study protocol for the duration of the study including scheduled clinic appointments.
8. Able and willing to provide written informed consent for study participation prior to performance of any study-related assessments.

Exclusion Criteria:

1. Subject has signs of or is diagnosed with Type 1 diabetes mellitus or latent autoimmune diabetes in adults.
2. History of hospitalizations or emergency room visits that would impact subject safety or data interpretation, including:

   * Poor glucose control in the 6 months prior to Screening (per investigator discretion) or
   * Any bariatric surgical procedures for weight loss.
3. History of significant change of body weight (> 10%) in the 3 months prior to Screening.
4. History of or active proliferative retinopathy or maculopathy within the 6 months before Screening or requiring acute treatment, or severe neuropathy.
5. History of previous gastrointestinal bleeding or ulceration within 3 months prior to Screening.
6. History of acute or chronic pancreatitis.
7. History of significant cardiovascular events defined as:

   * Myocardial infarction, coronary angioplasty or bypass grafts, valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accidents within 6 months prior to Screening.
   * Congestive heart failure defined as New York Heart Association (NYHA) Stages III and IV.
   * Uncontrolled hypertension defined as a systolic blood pressure > 160 mmHg and/or a diastolic blood pressure > 100 mmHg.
   * Symptomatic postural hypotension - The difference between supine blood pressure and standing blood pressure is 20 mmHg in systolic or 10 mmHg in diastolic with any symptom.
8. Evidence of uncorrected hypothyroidism or hyperthyroidism based on clinical evaluation and/or an abnormal thyroid stimulating hormone result as determined at Screening; subjects receiving dose-stable thyroid replacement therapy for at least 3 months prior to Screening will be allowed to participate in the study.
9. History of significant other major or unstable neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, or urological disorder that would impact subject safety or data interpretation.
10. History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening ( subjects with a history of treated cervical intraepithelial neoplasia will be allowed to participate in the study).
11. Active liver disease and/or significant abnormal liver function defined as aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN) and/or alanine aminotransferase (ALT) > 2.5 × ULN and/or total bilirubin > 2.0 mg/dL.
12. Positive blood screen for anti-hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), and human immunodeficiency (HIV) antibody.
13. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, ECG, or clinical laboratory assessments.
14. Long QT syndrome or prolongation of QTc interval (defined as QTc interval > 460 ms for males and > 480 ms for females).
15. The following medication exclusions apply:

    * Use of weight control treatment 3 months prior to Screening, including any medication with a labeled reference to weight loss or gain, herbal preparations, and over the counter medications.
    * Use of other anti-diabetic agents (except metformin) within 3 months prior to Screening (if the subject was previously treated with thiazolidinedione, he/she must have stopped this treatment at least 6 months before Screening).
    * Use of insulin within 12 months prior to Screening (the following cases can be included in this study: Insulin treatment during hospitalization, insulin treatment for a medical condition that did not require hospitalization [< 2 weeks treatment period], or insulin treatment for gestational diabetes).
16. Treatment with an investigational agent within the longest time frame of either 5 half lives or 30 days of initiating study drug.
17. Use of prohibited concomitant medications (further details about prohibited medication are provided in Section 5.8.1):

    * Current use of hyperglycemia-causing agents, hypoglycemia-causing agents, Class II and III antiarrhythmic agents (these agents will be allowed if they have been used for hypertension treatment), agents that reduce gastrointestinal motility, central nervous system stimulants (with the exception of caffeinated beverages), and niacin ≥ 1 g/day.
    * Current use of drugs with a narrow therapeutic index (eg, digoxin, lithium, phenytoin, theophylline, and warfarin).
    * Current use of drugs that are known to prolong the QT interval.
18. Known recreational substance use or psychiatric illness that, in the opinion of the Investigator, may impact the safety of the subject or the study objectives (eg, cannot comply with scheduled study visits).
19. History of drug abuse.
20. Women who are pregnant (confirmed by laboratory testing), nursing or are planning to become pregnant.
21. Subject is not willing to use an "effective" method of contraception during the course of the study. Sexually active male subjects are required to use a condom, abstain from intercourse, or previously undergone male sterilization. Male subjects should refrain from sperm donation for the purposes of conception for at least 90 days after their last dose of study drug. Females subjects must be surgically sterile (ie, hysterectomy or bilateral tubal ligation), postmenopausal, or for women of childbearing potential using a medically acceptable method of contraception (ie, intrauterine device, barrier methods with spermicide or abstinence). Female subjects of childbearing potential taking stable oral, implantable, or injectable contraceptives must additionally use a double-barrier method of contraception.
22. Subject has an FPG ≥ 270 mg/dL at the Screening visit.
23. Has a serum creatinine above (or creatinine clearance below) what is approved in the metformin product labeling in the respective country.
24. Known allergy or hypersensitivity to MLR-1023 or components of the formulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c between active treatment groups and placebo at Week 12 | 12 Weeks
  Change in HbA1c from Baseline to Week 12

SECONDARY OUTCOMES:
HbA1c of < 7.0% at Week 12 | 12 Weeks
  Proportion of Subjects with HbA1c of < 7.0% at Week 12
HbA1c of < 6.5% at Week 12 | 12 Weeks
  Proportion of Subjects with HbA1c of < 6.5% at Week 12
Changes in Fasting Plasma Glucose (FPG) from Baseline to Week 12 between active treatment groups and placebo | 12 Weeks
  Changes in FPG from Baseline to Week 12
Changes in fasting insulin, insulin sensitivities (HOMA IR) | 12 Weeks
  Changes in fasting insulin, insulin sensitivities (HOMA IR) from Baseline to Week 12
Changes in lipid profile (low density lipoprotein cholesterol [LDL-C], high density lipoprotein cholesterol [HDL-C], triglycerides) | 12 Weeks
  Changes in lipid profile (low density lipoprotein cholesterol [LDL-C], high density lipoprotein cholesterol [HDL-C], triglycerides) from Baseline to Week 12
Changes in Body Weight | 12 Weeks
  Changes in Body Weight from Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ramana Kuchibhatla, PhD, Study Director — Melior Pharmaceuticals, Inc.
Locations (1):
- National Research Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided